CLINICAL TRIAL: NCT02254135
Title: A Randomised, Single-blind, Placebo-controlled (Within Dose Groups) Study to Assess Safety, Tolerability and Pharmacokinetics of Single Rising Peroral Doses (400, 800, 1200 μg Free Cation) BEA 2180 BR in Healthy Male Volunteers
Brief Title: Study to Assess Safety, Tolerability and Pharmacokinetics of Single Rising Doses of BEA 2180 BR in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1205.20
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy

ARMS (2):
- BEA 2180 BR solution - rising dose (Experimental)
  Interventions: Drug: BEA 2180 BR - rising dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BEA 2180 BR - rising dose
  Arms: BEA 2180 BR solution - rising dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to investigate safety, tolerability, and pharmacokinetics of single rising peroral doses of BEA 2180 BR

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
2. Age ≥21 and ≤55 years
3. BMI ≥18.5 and <30 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including BP, PR, and ECG measurements) deviating from normal and of clinical relevance
2. Evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of relevant allergy/hypersensitivity (including allergy to the drug or its excipients) as judged clinically relevant by the investigator
8. Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to randomisation
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to enrolment in the study or during the study
10. Participation in another trial with an investigational drug within 30 days prior to randomisation
11. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
12. Inability to refrain from smoking on trial days as judged by the investigator
13. Alcohol abuse (regularly more than 40 g alcohol per day)
14. Drug abuse
15. Blood donation (more than 100 mL blood within 4 weeks prior to randomisation or during the trial)
16. Excessive physical activities within 1 week prior to randomisation or during the trial
17. Any laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of the study centre

    The following exclusion criteria are specific for this study due to the known class side effect profile of anticholinergic drugs:
19. History of hypersensitivity to tiotropium and/or related drugs of these classes
20. History of narrow-angle glaucoma
21. History of prostatic hyperplasia
22. History of bladder-neck obstruction

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-12; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects with abnormal findings in physical examination | up to 14 days after last procedure
Number of subjects with clinically significant changes in vital signs | up to 14 days after last procedure
  (Blood pressure (BP), pulse rate (PR), respiration rate (RR), oral body temperature)
Number of subjects with clinically significant changes in 12-lead electrocardiogram (ECG) | up to 14 days after last procedure
Number of subjects with abnormal changes in laboratory parameters | up to 14 days after last procedure
Number of subjects with adverse events | up to 14 days after last procedure
Assessment of tolerability by the investigator on a 4-point scale | 14 days after last procedure

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 48 h after drug administration
tmax (time from dosing to maximum measured concentration of the analyte in plasma) | up to 48 h after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 48 h after drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | up to 48 h after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 48 h after drug administration
λz (terminal rate constant in plasma) | up to 48 h after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 48 h after drug administration
MRTpo (mean residence time of the analyte in the body after peroral administration) | up to 48 h after drug administration
CL/F (clearance of the analyte in plasma after peroral administration) | up to 48 h after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following a peroral dose) | up to 48 h after drug administration
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | up to 48 h after drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 48 h after drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 48 h after drug administration